CLINICAL TRIAL: NCT06842160
Title: Photoplethysmography (PPG) Algorithm with Smartwatch in Evaluation of Atrial Fibrillation Burden After Catheter Ablation
Acronym: Polaris-AFCA
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KS2024101; KS2024101 (Other: Chengdu Xinjikang Technology Co., Ltd)
Record Dates: First submitted 2024-12-04; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial Fibrillation Burden、 Catheter Ablation; Photoplethysmography; Wearable devices.
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Electrocardiogram data、Photoplethysmography data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: intervention group — A smart electrocardiogram watch based on the PPG algorithm for monitoring atrial fibrillation load after catheter ablation.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a smart electrocardiogram watch based on the PPG algorithm in monitoring the atrial fibrillation burden of patients after catheter ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Atrial fibrillation patients diagnosed by electrocardiogram
2. Received catheter ablation procedure
3. Willing to use long-range electrocardiogram monitoring equipment

Exclusion Criteria:

1.Patients who are allergic to electronic devices or unable to wear watches

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have undergone catheter ablation for atrial fibrillation and meet age and health standards are able to use electrocardiographic watches for long-term monitoring
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2035-03-30 (Estimated); Study Completion 2036-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Stroke | March 30, 2025 to March 30, 2035
  The rate of stroke occurrences in the study population, measured separately for each participant. The unit of measure will be the frequency of events (e.g., number of strokes per participant).
Incidence of Heart Failure | March 30, 2025 to March 30, 2035
  The rate of heart failure occurrences in the study population, measured separately for each participant. The unit of measure will be the frequency of events (e.g., number of heart failure episodes per participant).
All-Cause Mortality Rate | March 30, 2025 to March 30, 2035
  The rate of all-cause mortality in the study population, measured separately for each participant. The unit of measure will be the frequency of events (e.g., number of deaths per participant).
Cardiovascular Mortality Rate | March 30, 2025 to March 30, 2035
  The rate of cardiovascular-related mortality in the study population, measured separately for each participant. The unit of measure will be the frequency of events (e.g., number of cardiovascular-related deaths per participant).
Rate of Rehospitalization | March 30, 2025 to March 30, 2035
  The rate of rehospitalization due to any medical cause in the study population. The unit of measure will be the frequency of events (e.g., number of rehospitalization events per participant).
Incidence of Bleeding Events | March 30, 2025 to March 30, 2035
  The rate of bleeding events (such as major or minor bleeding) in the study population. The unit of measure will be the frequency of events (e.g., number of bleeding events per participant).
Postoperative Atrial Fibrillation Burden | March 30, 2025 to March 30, 2035
  The frequency and severity of atrial fibrillation episodes observed in participants after a surgical procedure, measured using data collected by an intelligent heart rate monitoring watch utilizing a PPG algorithm. The unit of measure will be frequency of events (e.g., number of episodes per participant).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No